CLINICAL TRIAL: NCT04344509
Title: Microbial Etiology of Ventilator-associated Pneumonia (VAP) in COVID-19 Infected Patients
Brief Title: Microbial Etiology of Ventilator-associated Pneumonia in COVID-19 Infected Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PAVM COVID
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-04

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID19-positive patients
  Interventions: Other: Bacterial species isolated
- COVID19-negative patients
  Interventions: Other: Bacterial species isolated

INTERVENTIONS:
Other: Bacterial species isolated — in the respiratory specimen

SUMMARY:
National multicentric observational retrospective case-control study comparing the relative frequency of the various microorganisms responsible for VAP in patients infected or not by SARS-CoV-2 and their resistance to antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* All patients with microbiologically confirmed VAP with pulmonary samples collected from March 15 to April 15 in France.

Exclusion Criteria:

* All patients with microbiologically confirmed VAP with pulmonary samples collected from March 15 to April 15 in France.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with microbiologically confirmed VAP with pulmonary samples collected from March 15 to April 15 in France.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the microorganisms responsible for VAP among patients infected or not by the SARS-CoV-2 | 1 month

SECONDARY OUTCOMES:
Prevalence of multi-drug resistant bacteria responsible for VAP among patients infected or not by the SARS-CoV-2 | 1 month

IPD SHARING:
Plan to Share IPD: No